CLINICAL TRIAL: NCT02423772
Title: Pilot Study of Combined Treatment for Veterans With Chronic Pain & Opiate Misuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AT008398-01
Record Dates: First submitted 2015-04-09; First posted 2015-04-22 (Estimated); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-08

CONDITIONS: Chronic Pain; Problematic Opioid Use
MeSH Terms: conditions — Chronic Pain | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Treatment as usual, plus 12 weeks of group based intervention to improve functioning and decrease problematic effects of opioid use.
  Interventions: Behavioral: Acceptance and Commitment Therapy + Mindfulness-Based Relapse Prevention + Treatment as Usual (TAU)
- Treatment as Usual (No Intervention)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy + Mindfulness-Based Relapse Prevention + Treatment as Usual (TAU)
  Arms: Intervention

SUMMARY:
Chronic pain and misuse of opioids is a major public health problem, particularly in military veterans. The major goal of this project is to test the efficacy of an innovative behavioral treatment for chronic pain patients who are misusing prescription opiates. This project supports the strategic goals of National Center for Complementary and Integrative Health (NCCIH) and National Institute on Drug Abuse by examining a difficult and understudied problem with the ultimate goal of impacting scientific knowledge and human health.

DETAILED DESCRIPTION:
Opioid prescription in the treatment of chronic pain is frequent and carries a consequent risk of poor treatment outcome, as well as higher morbidity and mortality in a clinically significant number of patients, particularly those who meet criteria for opioid dependence. Despite the alarming increases (140% increase from 1992 to 2003) in prescription opiate misuse, abuse, and dependence nationally in the United States, there are few treatment options available that target both pain-related interference and opioid dependence among patients with chronic pain. In military veterans, this issue is of particular importance as numerous reports indicate increasing use of opioids in the treatment of chronic pain, as well as increasing opioid-related problems, specifically in those who served in the Iraq and Afghanistan theatres [Operation Enduring Freedom (OEF), Operation Iraqi Freedom (OIF), and Operation New Dawn (OND)]. To date, there are no evidenced-based treatment options which aim to both maximize effective functioning in Veterans with chronic pain while simultaneously addressing problematic opioid use. The overall aim of the present study will be to determine the feasibility of an integrated psychosocial treatment in veterans with chronic pain, who also have evidence of opioid-related misuse. To examine this aim, the investigators will utilize a randomized design to assess the feasibility of integrating two empirically supported interventions: Acceptance and Commitment Therapy for chronic pain and Mindfulness Based Relapse Prevention for substance use and misuse. Feasibility will be assessed by examining rates of recruitment and retention of participants through a six month follow-up. In addition, the investigators will evaluate progress within-treatment on specific therapy targets to aid in the identification of potential treatment mechanisms. The results of this study will directly inform treatment of chronic pain patients and represents a significant advance in the growing and understudied problem of opiate misuse among chronic pain patients. In addition to addressing the question of whether the treatment is feasible, it will further examine issues of treatment mechanisms to better inform the design of a randomized and controlled trial assessing treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-65 years old
* Diagnosis of chronic pain condition
* Pain severity over the past seven days of four or greater on a 0-10 scale
* Prescribed opioids for the treatment of chronic pain for the past 90 days or longer
* Ability to read written English

Exclusion Criteria:

* Meet diagnostic criteria for current substance abuse/dependence on a drug other than opioids
* Meet diagnostic criteria for a current or past DSM diagnosis of schizophrenia, delusional disorder, psychotic or dissociative disorders,
* Currently prescribed medications for opioid addiction (e.g., Buprenorphine/Naloxone/Suboxone).
* History of suicide attempts or inpatient hospitalization for risk of suicide in the past six month. In addition, we will screen for significant suicidal

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Raymond G. Murphy VA Medical Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pielech M, Kruger E, Rivers WE, Snow HE, Vowles KE. Receipt of multiple outpatient opioid prescriptions is associated with increased risk of adverse outcomes in youth: opioid prescribing trends, individual characteristics, and outcomes from 2005 to 2016. Pain. 2020 Jun;161(6):1297-1310. doi: 10.1097/j.pain.0000000000001812. PMID 31977934
- [Background] Witkiewitz K, Votaw VR, Vowles KE, Kranzler HR. Opioid Misuse as a Predictor of Alcohol Treatment Outcomes in the COMBINE Study: Mediation by Medication Adherence. Alcohol Clin Exp Res. 2018 Jul;42(7):1249-1259. doi: 10.1111/acer.13772. Epub 2018 Jun 9. PMID 29873089
- [Background] Vowles KE, Bailey RW, McEntee ML, Pielech M, Edwards KA, Bolling LA, Rivers WE. Using Analgesics for Emotional Modulation is Associated With Increased Distress, Depression, and Risk of Opioid and Alcohol Misuse: Initial Evaluation and Component Analysis of the Reasons for Analgesic Use Measure (RAUM). Clin J Pain. 2018 Oct;34(10):975-982. doi: 10.1097/AJP.0000000000000621. PMID 29697475
- [Background] Witkiewitz K, Vowles KE. Alcohol and Opioid Use, Co-Use, and Chronic Pain in the Context of the Opioid Epidemic: A Critical Review. Alcohol Clin Exp Res. 2018 Mar;42(3):478-488. doi: 10.1111/acer.13594. Epub 2018 Feb 6. PMID 29314075
- [Background] Bailey RW, Vowles KE. Using Screening Tests to Predict Aberrant Use of Opioids in Chronic Pain Patients: Caveat Emptor. J Pain. 2017 Dec;18(12):1427-1436. doi: 10.1016/j.jpain.2017.06.004. Epub 2017 Jun 29. PMID 28669863
- [Background] Pielech M, Vowles KE, Wicksell R. Acceptance and Commitment Therapy for Pediatric Chronic Pain: Theory and Application. Children (Basel). 2017 Jan 30;4(2):10. doi: 10.3390/children4020010. PMID 28146108
- [Background] Witkiewitz K, McCallion E, Vowles KE, Kirouac M, Frohe T, Maisto SA, Hodgson R, Heather N. Association between physical pain and alcohol treatment outcomes: The mediating role of negative affect. J Consult Clin Psychol. 2015 Dec;83(6):1044-57. doi: 10.1037/ccp0000033. Epub 2015 Jun 22. PMID 26098375
- [Background] Witkiewitz K, Vowles KE, McCallion E, Frohe T, Kirouac M, Maisto SA. Pain as a predictor of heavy drinking and any drinking lapses in the COMBINE study and the UK Alcohol Treatment Trial. Addiction. 2015 Aug;110(8):1262-71. doi: 10.1111/add.12964. Epub 2015 Jun 3. PMID 25919978
- [Result] Vowles KE, Witkiewitz K, Cusack KJ, Gilliam WP, Cardon KE, Bowen S, Edwards KA, McEntee ML, Bailey RW. Integrated Behavioral Treatment for Veterans With Co-Morbid Chronic Pain and Hazardous Opioid Use: A Randomized Controlled Pilot Trial. J Pain. 2020 Jul-Aug;21(7-8):798-807. doi: 10.1016/j.jpain.2019.11.007. Epub 2019 Nov 21. PMID 31760109

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Treatment as usual, plus 12 weeks of group based intervention to improve functioning and decrease problematic effects of opioid use.
  Acceptance and Commitment Therapy + Mindfulness-Based Relapse Prevention + Treatment as Usual (TAU).
  Assessment at randomization, post-intervention (12 weeks post randomization), and six month follow-up (9 months post randomization; 6 months after end of intervention).
- Treatment as Usual: Physician directed care through a VA co-occurring disorders clinic that primarily provided medical oversight of opioid prescription and directed patients to other necessary pain interventions.
  Assessment at randomization, post-intervention (12 weeks post randomization), and six month follow-up (9 months post randomization; 6 months after end of intervention).
Period: Overall Study
Arm/Group | Intervention | Treatment as Usual
Started | 17 | 18
Received Allocated Intervention | 15 | 13
Completed ("Completed" defined as provided 6 month follow-up data.) | 12 | 10
Not Completed | 5 | 8
Not completed — Lost to Follow-up | 3 | 3
Not completed — Did not begin intervention | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Treatment as Usual | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.3 (11.6) | 53.3 (8.6) | 50.5 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 14 | 16 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 13 | 11 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 7 | 18
  More than one race | 3 | 7 | 10
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) - Pain Behavior
Description: The PROMIS pain behavior (PROMIS short form v1.1 7a) measures self-reported frequency of verbal and nonverbal behaviors indicating that one is experiencing pain. It consists of 7 items with scores ranging from 7 to 35 with higher scores indicating more frequent pain behavior.
Time Frame: Change from baseline (i.e., the beginning of the intervention) in Pain behavior, as measured by PROMIS at 9 months post randomization (6 months post end of intervention period).
Population: Per protocol analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Treatment as Usual
Number analyzed (Participants) | 17 | 18
units on a scale
  Baseline | 66.7 (6.6) | 66.0 (6.6)
  6 month follow-up | 64.3 (9.2) | 66.8 (8.0)

2. Primary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) - Pain Interference
Description: The PROMIS pain interference Short Form 8a assesses the impact of pain on important aspects of social, physical, cognitive, and recreational activities. It consists of 8 items and scores range from 8 to 40 with higher scores indicating greater pain interference.
Time Frame: as for outcome 1
Population: Per protocol analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Treatment as Usual
Number analyzed (Participants) | 17 | 18
units on a scale
  Baseline | 66.7 (6.6) | 65.2 (6.8)
  6 month follow-up | 64.3 (9.2) | 70.1 (4.9)

3. Primary Outcome: Current Opioid Misuse Measure (COMM)
Description: Total Score of the COMM was used. The COMM is a 17-item measure designed to aid in the identification of opioid misuse. Scores range from 0 to 68 with higher scores indicating greater risk of misuse.
Time Frame: Change from baseline (i.e., the beginning of the intervention) in Pain behavior, as measured by PROMIS at 9 months post randomization (6 months
Population: Per protocol analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Treatment as Usual
Number analyzed (Participants) | 17 | 18
units on a scale
  Baseline | 16.2 (8.8) | 17.4 (7.8)
  6 month follow-up | 10.6 (6.5) | 16.1 (8.5)

ADVERSE EVENTS:
Time Frame: Study period was (9 months) to include the three month intervention period and six month post-intervention follow-up period. Specific dates of the study period was from 21 April 2015 through 13 March 2018.
Description: The PI of the study (Dr. Vowles) reported all adverse events to the IRB of record. For any adverse events, a course of remediation was planned to be proposed (e.g., in the event of a protocol violation, safeguards will be put in place to decrease the probability of repeated violation) to the IRB, although the IRB itself took responsibility to approve/disapprove the remediation. All AE's reported within five days. A Data Safety Monitoring Board met at least yearly to review all such events.
Arm/Group | Intervention | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 0/17 | 0/18

LIMITATIONS AND CAVEATS:
This was a pilot trial intended to test feasibility and a preliminary test of efficacy. Sample size was small, which places limits on generalizability and power. TAU did not include a active psychotherapy comparator. The study was under-recruited, which indicates poorer than expected feasibility. Finally, we did not assess therapist competency in treatment delivery; we did assess adherence to the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-22): https://cdn.clinicaltrials.gov/large-docs/72/NCT02423772/Prot_SAP_000.pdf